CLINICAL TRIAL: NCT07369908
Title: The Modulatory Effects of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) on Anxiety Responses and Emotional Regulation
Brief Title: The Effects of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) on Anxiety Responses and Emotional Regulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-97
Record Dates: First submitted 2025-09-29; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-09

CONDITIONS: Healthy Male and Female Volunteers
Keywords: taVNS; anxiety; emotional regulation; high-trait anxiety
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experiment and high trait anxiety group (Experimental): male and female subjects with high trait anxiety and experimental treatment
  Interventions: Device: taVNS on tragus of subjects with high trait anxiety
- Sham control and high trait anxiety group (Sham Comparator): male and female subjects with high trait anxiety and sham treatment
  Interventions: Device: taVNS on earlobe of subjects with high trait anxiety
- Experiment and no high trait anxiety group (Experimental): male and female subjects with no high trait anxiety and experimental treatment
  Interventions: Device: taVNS on tragus of subjects with no high trait anxiety
- Sham control and no high trait anxiety group (Sham Comparator): male and female subjects with no high trait anxiety and sham treatment
  Interventions: Device: taVNS on earlobe of subjects with no high trait anxiety

INTERVENTIONS:
Device: taVNS on tragus of subjects with high trait anxiety — 15 minutes taVNS on tragus
  Arms: Experiment and high trait anxiety group
Device: taVNS on earlobe of subjects with high trait anxiety — 15 minutes taVNS on earlobe
  Arms: Sham control and high trait anxiety group
Device: taVNS on tragus of subjects with no high trait anxiety — 15 minutes taVNS on tragus
  Arms: Experiment and no high trait anxiety group
Device: taVNS on earlobe of subjects with no high trait anxiety — 15 minutes taVNS on earlobe
  Arms: Sham control and no high trait anxiety group

SUMMARY:
The main aim of this study is to investigate whether transcutaneous auricular vagus nerve stimulation (taVNS) can reduce anxiety and have an effect on emotional regulations

DETAILED DESCRIPTION:
Transcutaneous auricular vagus nerve stimulation (taVNS) is a non-invasive method for modulating vagal nerve function and has shown potential efficacy in alleviating anxiety symptoms and improving emotional regulation. But the neural mechanisms of how taVNS affects anxiety and emotional regulation remain unclear. Therefore, we focus on this question by combining behavioral meausres, skin conductance response, heart rate variability and fMRI in this study. A participant-blinded, sham-controlled, between-subject design is employed in this study. In a randomised order, a total of 140 healthy males and females with or without high trait anxiety are recruited and receive the stimulation of taVNS on their tragus (experimental group) or earlobe (sham control group). After the participants arrive at the laboratory, they first complete a roughly 30-minute personality trait questionnaire and prepare for the experiment. Then, they undergo a 7-minute resting-state fMRI scan, followed by a 15-minute taVNS session. Next, they complete a 7-minute resting-state scan and a 60-minute task-based scan (a modified emotional regulation task). During the entire procedure, saliva samples will be collected three times for subsequent physiological hormone analyses, and participants' skin conductance and electrocardiogram data will also be recorded. During the modified emotional regulation task, subjects are instructed to regulate their emotional responses to negative pictures (high vs. low intensity) using reinterpretation/distance strategies or to only look these pictures. We also record subjects' rating scores on their anxiety levels during these conditions ("reinterpretation" vs. "distance" vs. "look") and successful usage of emotional regulation strategies. Questionnaire scores including State-Trait Anxiety Inventory, Beck Depression Inventory II, Beck Anxiety Inventory, Autism Spectrum Quotient, Toronto Alexithymia Scale, Social Responsiveness Scale, Emotion Regulation Questionnaire, Cognitive Emotion Regulation Questionnaire, Multidimensional Assessment of Interoceptive Awareness, Positive and Negative Affect Schedule will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders.

Exclusion Criteria:

* History of head injury.
* Medical or psychiatric illness.
* Subjects take a certain drug for a long period of time.
* Subjects have metal implants in their bodies.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-04-16 (Estimated)

PRIMARY OUTCOMES:
Brain activity patterns in response to negative pictures during emotional regulation | 60 minutes
  Subjects will receive task-based fMRI scanning (i.e., the modified emotional regulation task) after taVNS and two resting-state fMRI scanning sessions. We will examine these brain response patterns in the modified emotional regulation task via both the conventional univariate analysis and the machine learning-based multivariate pattern analysis.
Resting-state functional conetivity changes | 15 minutes
  Subjects will receive resting-state fMRI scanning twice before and after taVNS. We will examine resting-state functional conetivity changes induced by taVNS via examining functional conetivity differences between pre- and post-taVNS sessions.
Behavioral indices in the task | 60 minutes
  Anxiety and success ratings after each regulation trial are recorded in the task. Subjects are instructed to rate their anxiety and success levels using a 9-point Likert scale within 4 seconds (1 = not at all, 9 = very anxious or successful)

SECONDARY OUTCOMES:
Skin conductance responses (SCR) in the emotional regulation task during fMRI scanning | 60 minutes
  Skin Conductance Response (SCR) data in response to negative pictures while using different regulation strategies are recorded in the emotional regulation task.
HRV in resting-state fMRI and emotional regulation task | 75 minutes during scanning
  Heart beat variability (HRV) data are recorded in resting-state fMRI and emotional regulation task.
Saliva samples analysis | Three time points: pre-taVNS (baseline, 0 minute), immediate post-taVNS (60 minutes post-taVNS), and the end of experiment (70 minutes post-scanning).
  Saliva samples will be collected three times for subsequent physiological hormone analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shuxia Yao, Dr, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China (UESTC), Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No